CLINICAL TRIAL: NCT02695680
Title: Modeling Respiration-induced Motion and Deformation of Tumors and Thoracic Organs for Personalized Motion Management in Lung SBRT
Brief Title: Lung SBRT Motion Management (GCC 1619)
Status: Terminated | Type: Observational
Why Stopped: Funding for this study is over and the PI has request closure.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00068540
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; SBRT; Motion Management
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung SBRT: Respiratory motion causes significant geometric and dosimetric errors in the administration of lung stereotactic radiotherapy (SBRT). The purpose of this study is to create and validate patient-specific motion models of the thoracic anatomy with high spatial and temporal resolution. These models will be used to develop novel four-dimensional (4D=3D+time) techniques for radiotherapy treatment planning and real-time motion-adaptive dose delivery.

SUMMARY:
Real-time optical surface monitoring data will be acquired from 44 human patients with primary or metastatic lung lesions during and after their 4DCT scan (standard-of-care at our institution). A patient-specific 4D model will be developed using the raw 4DCT projections time-correlated with real-time surface monitoring. In addition, before delivering each dose fraction (3 - 5 for lung SBRT), we will acquire three 15s kV fluoroscopic image acquisitions, time-correlated with optical surface monitoring. The acquisitions will be distributed over three well-spaced beam angles, e.g., every 4th angle for a 12-field plan.

DETAILED DESCRIPTION:
Surface monitoring procedure -The procedure is expected to last approximately 15 minutes after the end of the 4DCT scan, which is the standard-of-care for lung SBRT treatments at our institution. The procedure will consist of real-time surface tracking using the VisionRT system of the thoracic and/or abdominal region. Continuous audiovisual contact will be maintained with the subject during scanning. Each individual will be informed that they can stop the procedure at any point.

Fluoroscopic imaging procedure - Fluoroscopic imaging will be performed in the treatment room with the patient lying in treatment position. Three 15s acquisitions will be performed under free breathing conditions, each from a different beam angle, using the on-board kV imager. Audiovisual contact will be maintained at all times with the patient.

Data collection and management: An ID number will be assigned to each separate patient, and the correlation between ID number and patient name and medical record number will be kept in a password-protected file in Dr. Amit Sawant's office. The database of information extracted from the medical record and radiation treatment records for each patient will be stored in an Excel file on a computer with password protection. All image data will be de-identified by Dr. Sawant before his research team analyzes them.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible disease(s)/stage(s) - Patients with primary or metastatic lung lesions to be treated using stereotactic body radiotherapy (SBRT) will be eligible for this study.
2. Allowable type and amount of prior therapy - Any types and amounts of prior therapy will be allowed for this study.
3. Age restriction and/or gender/ethnic restrictions - Patients must be greater than or equal to 18 years of age. There are no gender or ethnic restrictions.
4. Life expectancy restrictions - None.
5. ECOG or Karnofsky Performance Status - Karnofsky performance status of 50 or greater
6. Requirements for organ and marrow function - None.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Tumor motion > 5 mm, maximum GTV dimension < 50 mm - per guidelines established by the AAPM Task Group 7612 and RTOG 0236.13

Exclusion Criteria:

1. Children (age <18)
2. Women who are pregnant or trying to get pregnant
3. Pain in supine position
4. Karnofsky performance status < 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or metastatic lung lesions
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who demonstrate significant motion movement during radiation therapy. | 1.5 years
  Develop novel Four-dimensional (4D=3D+time) techniques for radiotherapy treatment planning and real-time motion-adaptive dose delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sawant, PhD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - Ummc Msgcc, Baltimore, Maryland
  - Upper Chesapeake Health, Bel Air, Maryland

IPD SHARING:
Plan to Share IPD: No